CLINICAL TRIAL: NCT02302326
Title: Involvement of Reticulum Endoplasmic Stress in the Physiopathology of Polycystic Ovary Syndrome: Possible Therapeutic Implications of Insulin Sensitizers.
Brief Title: Involvement of Reticulum Endoplasmic Stress in the Physiopathology of Polycystic Ovary Syndrome
Acronym: PI12/1984
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Antonio Hernandez Mijares, PhD, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHM-MET-2013-01
Record Dates: First submitted 2014-10-29; First posted 2014-11-27 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: reticulum endoplasmic stress; Polycystic Ovary Syndrome; mitochondrial function; insulin resistance; inflammation; myoinositol; metformin; oxidative stress
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Inflammation | interventions — Metformin; Inositol; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Experimental): PCOS women began treatment with ER 500 mg metformin per day, and the dose was increased to 1000 mg after 2 weeks, and to 1700 mg/d after a further 2 weeks, and was maintained at this dose for a total of 12 weeks.
  Interventions: Drug: Metformin
- Myo-inositol + folic acid (Experimental): PCOS women received a dietary supplement (Ovusitol® : 4 g myo-inositol plus 400 micrograms of folic acid) for 12 weeks
  Interventions: Dietary Supplement: Myo-inositol + folic acid
- Healthy women (No Intervention): Healthy untreated women adjusted for age and body mass index

INTERVENTIONS:
Drug: Metformin — Dose: metformin (1700 mg / day) for 12 weeks
  Arms: Metformin
Dietary Supplement: Myo-inositol + folic acid — Dose: Ovusitol® (4 g myo-inositol plus 400 micrograms of folic acid/day) for 12 weeks
  Arms: Myo-inositol + folic acid

SUMMARY:
The main objective of the present project is to evaluate the relevance of reticulum stress in the pathogenesis of polycystic ovary syndrome (PCOS), focusing particularly on the underlying mechanisms of insulin resistance, which is the origin of metabolic comorbidities. Furthermore, the investigators will assess the potential of insulin sensitizers as a treatment to control endoplasmic reticulum stress markers in PCOS patients.

DETAILED DESCRIPTION:
To do this, the investigators will evaluate anthropometric, biochemical and hormone parameters, lipid profile and cardiovascular risk markers (using enzymatic and biochemical techniques, nephelometry, enzyme-linked immunosorbent assay, radioimmunoassay), and markers of endoplasmic reticulum stress and the insulin pathway and inflammatory and apoptotic parameters (by means of Western blot, Real Time- Polymerase Chain Reaction (RT-PCR), Luminex® xMAP® Technology ) in patients with and without PCOS. The investigators' second objective is to evaluate (using the abovementioned methodology) the efficacy of different insulin sensitizers (myoinositol and metformin) administered to PCOS patients during a 3-month period after which the investigators will analyze different parameters of oxidative stress and mitochondrial function (using Clark electrode and fluorometric techniques).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS using the Rotterdam criteria
* Women of reproductive age

Exclusion Criteria:

* Organic, malignant, haematological, infectious or inflammatory disease
* History of ischaemic heart disease (stroke or thromboembolism)
* Diabetes mellitus,
* Secondary causes of obesity (hypothyroidism, Cushing's syndrome)
* Severe hypertension.
* Smoking or alcohol habit

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in markers of endoplasmic reticulum stress in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Markers of endoplasmic reticulum stress (78-kDa glucose-regulated protein (GRP78), ubiquitous translation initiation factor 2α (eIF2α), double-stranded RNA-activated protein kinase (PERK), inositol requiring enzyme 1 (IRE1α), X-box binding protein 1 (XBP-1)) were assessed by Western Blot and Real Time- Polymerase Chain Reaction (RT-PCR) in polymorphonuclear cells
Changes in markers of the insulin pathway in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Markers of the insulin pathway (c-Jun N-terminal kinase (JNK), insulin receptor substrate (IRS)) were assessed by Western Blot and Real Time- Polymerase Chain Reaction (RT-PCR) in polymorphonuclear cells
Changes in inflammatory parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Inflammatory parameters (nuclear factor κB (NF-κB), interleukin-6 (IL6), tumor necrosis factor α (TNFα)) were assessed by Western Blot, Real Time- Polymerase Chain Reaction (RT-PCR), or Luminex® xMAP® Technology in polymorphonuclear cells and serum
Changes in apoptotic parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Apoptotic parameters (transcription factor C/EBP homologous protein (CHOP) and caspase 12) were assessed by Western Blot and Real Time- Polymerase Chain Reaction (RT-PCR) in polymorphonuclear cells

SECONDARY OUTCOMES:
Changes in anthropometric parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Anthropometric (weight, height, body mass index and waist) and blood pressure parameters were evaluated
Changes in biochemical parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Glucose levels were measured using enzymatic techniques. Insulin was measured by an enzymatic luminescence technique. IR was calculated by homeostasis model assessment (HOMA). Total cholesterol and triglycerides were measured by employing enzymatic assays, and high density lipoprotein cholesterol (HDLc) concentrations were recorded with an autoanalyser using a direct method. Low-density lipoprotein cholesterol (LDLc) concentration was calculated using the Friedewald method. Luteinizing hormone (LH), follicle stimulating hormone (FSH) and testosterone were measured by specific radioimmunoassays. Dehydroepiandrosterone-sulfate (DHEAS), sex hormone-binding globulin (SHBG), androstenedione and testosterone were measured by specific chemiluminescence techniques. High-sensitive C-reactive protein (hsCRP) was quantified by a latex-enhanced immunonephelometric assay
Changes in mitochondrial function parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Oxidative stress markers ( mitochondrial oxygen (O2) consumption, membrane potential, glutathione, reactive oxygen species (ROS) and hydrogen peroxide levels, mitochondrial mass) were assessed by Clark electrode and fluorometric techniques
Changes in endothelial function parameters in controls and pcos women before and after metformin/Myo-inositol + folic acid administration | 3 months
  Interactions between leukocytes and human umbilical vein endothelial cells were evaluated by flow chamber microscopy (leukocyte rolling velocity, leukocyte rolling flux and leukocyte adhesion). The vascular cell adhesion molecule 1 (VCAM-1), Intercellular adhesion molecule 1 (ICAM-1) and E-selectin were evaluated in serum by Luminex® 200 flow analyzer system

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernández, Phd, MD, Principal Investigator — FISABIO - University Hospital Dr Peset
Locations (1):
- Antonio Hernández, Valencia, Spain

REFERENCES:
- [Background] Hernandez-Mijares A, Banuls C, Gomez-Balaguer M, Bergoglio M, Victor VM, Rocha M. Influence of obesity on atherogenic dyslipidemia in women with polycystic ovary syndrome. Eur J Clin Invest. 2013 Jun;43(6):549-56. doi: 10.1111/eci.12080. Epub 2013 Mar 26. PMID 23528141
- [Background] Victor VM, Rocha M, Banuls C, Alvarez A, de Pablo C, Sanchez-Serrano M, Gomez M, Hernandez-Mijares A. Induction of oxidative stress and human leukocyte/endothelial cell interactions in polycystic ovary syndrome patients with insulin resistance. J Clin Endocrinol Metab. 2011 Oct;96(10):3115-22. doi: 10.1210/jc.2011-0651. Epub 2011 Jul 21. PMID 21778215
- [Background] Victor VM, Rocha M, Banuls C, Sanchez-Serrano M, Sola E, Gomez M, Hernandez-Mijares A. Mitochondrial complex I impairment in leukocytes from polycystic ovary syndrome patients with insulin resistance. J Clin Endocrinol Metab. 2009 Sep;94(9):3505-12. doi: 10.1210/jc.2009-0466. Epub 2009 Jun 30. PMID 19567514